CLINICAL TRIAL: NCT04153448
Title: Comparison of Sit-to-stand Test With Six-minute Walk Test in Bronchiectasis and Healthy Children
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Melih Zeren, Assistant Professor, Bezmialem Vakif University
Other Study IDs: bvumzeren04
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; Exercise capacity; Six-minute walk test; Sit-to-stand test
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bronchiectasis: Children with bronchiectasis
  Interventions: Other: Measurement of functional capacity
- Healthy Controls: Age-matched healthy volunteers
  Interventions: Other: Measurement of functional capacity

INTERVENTIONS:
Other: Measurement of functional capacity — Functional capacity of participants will be measured with six-minute walk test and sit-to-stand test

SUMMARY:
Children with bronchiectasis and age-matched healthy controls will be evaluated with sit-to-stand test and six-minute walk test and utilization of STST in determining functional capacity will be investigated.

DETAILED DESCRIPTION:
Bronchiectasis (BE) is a chronic condition which is characterized by the permanent abnormal widening of the bronchi as a result of repetitive airway infections and inflammation. Disabling cough and shortness of breath, excess mucus production, progressive airway obstruction and loss of skeletal muscle mass are the primary factors that impairs exercise tolerance in BE patients. Imaging modalities and pulmonary function test are insufficient to determine disease burden or the prognosis thus it is stated that exercise tolerance and quality of life should also be evaluated in these patients.

Exercise tolerance can be evaluated using cardiopulmonary exercise test by directly measuring oxygen consumption but the field tests such as six-minute walk test (6MWT), shuttle walk test or stair climbing tests also provides reliable data on exercise tolerance by measuring functional capacity. Among field tests, 6MWT is the most commonly used test for evaluating functional capacity in cardiopulmonary patients. Although 6MWT is easy to apply and does not require any special equipment, it still requires a 30-m long corridor and a total testing time of approx. 20 minutes considering the pre- and post-test resting periods which may impair its feasibility in some clinical settings.

Sit-to-stand test (STST) is firstly developed for older population to measure mobility related function and physical performance. Today, it is widely used in various populations including cardiopulmonary diseases such as cystic fibrosis, chronic obstructive pulmonary disease and heart failure. The investigator's aim in this study is to investigate whether STST is utilizable for evaluating functional capacity in children with BE.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-cystic fibrosis bronchiectasis

Exclusion Criteria:

* Hospitalization history in past month
* Diagnosis of other chronic pediatric diseases which may impair exercise tolerance such as cerebral palsy or neuromuscular disease
* Candidates for lung transplantation or history of lung transplantation

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children diagnosed with non-cystic fibrosis bronchiectasis and age matched healthy volunteers who do not have any diagnosed chronic diseases
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Six-minute walk test distance | 15 minutes
  Distance walked in six minutes will be recorded. Test will be conducted according to the guideline of American Thoracic Society (ATS).

SECONDARY OUTCOMES:
Number of repetitions in sit-to-stand test | 1 Minute
  Participants will be asked to perform sit-to-stand maneuver as fast as possible for 30 seconds and the number of completed repetitions will be recorded.
Forced Vital Capacity (FVC) | 5 minutes
  FVC will be measured using basic spirometry and expressed as the percentage of the predicted value according to the guideline of European Respiratory Society (ERS)
Forced Expiratory Volume in 1 second (FEV1) | 5 minutes
  FEV1 will be measured using basic spirometry and expressed as the percentage of the predicted value according to the guideline of European Respiratory Society (ERS)
Peak Expiratory Flow (PEF) | 5 minutes
  PEF will be measured using basic spirometry and expressed as the percentage of the predicted value according to the guideline of European Respiratory Society (ERS)
M. Quadriceps strength | 3 minutes
  Isometric M. Quadriceps strength will be measured using electronic hand held dynamometer in sitting position.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No